CLINICAL TRIAL: NCT06690866
Title: Negative Emotionality in Relation to Epigenetics of Estrogen Signaling During Puberty
Brief Title: Negative Emotionality and Epigenetics During Puberty
Status: Recruiting | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: University Hospital Tuebingen (Other); Uppsala University (Other); German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRTG_P01
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Puberty; Healthy; Stress
Keywords: Stress reactivity; DNA methylation; fMRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, saliva and hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-pubertal girls (children): 8-10 years of girls having pubertal stage 1
  Interventions: Behavioral: Stress
- Post-pubertal girls (adolescents): 15-17 years of girls having pubertal stage 5
  Interventions: Behavioral: Stress

INTERVENTIONS:
Behavioral: Stress — Montreal Imaging Stress Task is a stress paradigm in the scanner to examine neuronal correlates of acute psychosocial stress.

SUMMARY:
Pubertal transition leads to enduring neuroendocrine changes along with changes in the epigenome. The prevalence of psychiatric disorders significantly increases in females compared to males after puberty. There is likely to be an interaction between epigenetics, hormones and neurophysiological processes during puberty, leading to the increased prevalence of mental disorders in females. This study aims to shed light on these interactions underlying the emerging sex differences after puberty. Specifically, it seeks to investigate the epigenetic modifications and subsequent changes in gene expression during the pubertal transition and their association with negative emotionality (e.g., acute stress response and depressive symptoms) at molecular, neuronal, subjective and physiological levels.

DETAILED DESCRIPTION:
In order to investigate epigenetic and neuroimaging correlates of negative emotionality in pubertal girls, the study employs a cross-sectional design, enrolling 50 pre-pubescent girls (8-10 years) and 50 post-pubescent girls (15-17 years) as healthy participants. Comprehensive data will be collected using self- and parent-report questionnaires on pubertal status, prenatal complications, adverse life events, stress and coping mechanisms, mood and anxiety symptoms, gender identity, and reproductive health. To delve into the neuronal correlates of stress, participants will undergo (f)MRI and MIST. Additionally, physiological stress responses will be assessed through heart rate and skin conductance measurements. Participants will provide blood, saliva, and hair samples for hormone, methylation and expression analysis. DNA methylation analysis will be performed on whole blood and saliva samples using pyrosequencing, focusing on genes that are responsive to estrogen and genes involved in estrogen signaling, based on the previous literature reporting an overrepresentation of estrogen-responsive genes among the differentially methylated sites across the entire genome in girls during puberty. The effects of methylation on gene expression will be measured using reverse transcription real-time PCR. Cortisol levels will be assessed from saliva collected six times during MIST to evaluate the acute stress response and from hair to assess chronic stress. Sex steroids such as estrogen and progesterone from blood will be analyzed using LC-MS/MS. The study aims to provide insights into the intricate relationship between epigenetic modifications, gene expression and negative emotionality (e.g., stress reactivity and internalizing symptoms) during puberty in girls.

ELIGIBILITY:
Inclusion Criteria:

* healthy girls
* aged between 8-10 and having pubertal stage 1 or between 15-17 and having pubertal stage 5
* normal body mass index according to age (between 5th and 85th percentile)
* non-smoking
* German language fluency
* Attending age-appropriate schools

Exclusion Criteria:

* neurological or psychiatric disease
* medical problems such as hormonal, metabolic, developmental or chronic diseases (e.g., congenital disorders, precocious puberty, polycystic ovarian syndrome, diabetes or congestive heart failure)
* any kind of hormonal, pharmacological or psychotropic treatment in the last three months
* engaging in competitive/extreme sports

Additional exclusion criteria for MRI:

* People with non-removable metal objects on or in the body
* Tattoos (if not MRI-incompatible according to expert guidelines)
* Pathological hearing or increased sensitivity to loud noises
* Claustrophobia
* Surgery less than three months ago
* Moderate or severe head injury

Ages: 8 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pubescent girls between 8 and 17 years of age living and schooling in Tübingen and surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
DNA methylation differences between pre- and post-pubertal girls in candidate genes | Measured once after MRI measurement (approximately 30 minutes).
  DNA methylation (DNAm) leves in genes involved in estrogen signaling and neuronal estrogen responsive genes in blood and saliva
Correlation between DNA methylation and neuronal activity during acute stress | Measured once: 3 runs of MIST lasting 20 minutes in total.
  Neuronal activity during acute stress is determined by the contrast differences between stress and control conditions assessed with task-based fMRI, Montreal Imaging Stress Task (MIST). The correlation between neuronal activity and DNA methylation. Comparing pre- and post-pubescent girls.
The mediating role of sex steroids in DNA methlation and negative emotionality | Measured once for each part: 20 minutes for MIST, 30 minutes for blood and saliva collection, and 1 hour for questionnaires
  The mediating effect of estradiol, progesterone, testosterone and allopregnanolone levels in blood on the correlation between DNA methylation and indicators of negative emotionality (e.g., neuronal activity during stress (MIST task) and mood symptoms). Comparing pre- and post-pubescent girls

SECONDARY OUTCOMES:
Correlation between DNA methylation and gene expression in candidate genes | Measured once after MRI measurement (approximately 30 minutes)
  The expression levels of genes involved in estrogen signaling and neuronal estrogen responsive genes in blood and saliva with RT-PCR. Correlation between DNA methlaytion and expression.
Correlation between DNA methylation and HPA-axis response | Measured six times: 1 hour before MIST(1), just before(1) and after(1) MIST, and three times more in 20-minute intervals after MIST. Each saliva collection lasts approx. 2 minutes.
  Cortisol levels from saliva samples collected before and after MIST. Correlation between area under the curve (AUC) for cortisol and DNA methylation. Is there a mediating role of DNA methylation on the correlation between HPA-axis reactivity and negative emotionality (e.g., internalizing symptoms and stress processing)? Comparing pre- and post-pubescent girls.
Correlation between DNA methylation and subjective stress response | Measured six times: 1 hour before MIST(1), just before(1) and after(1) MIST, and three times more in 20-minute intervals after MIST. Each rating takes approx. 10 minutes.
  Correlation between emotional ratings and stress levels assessed with each saliva sample before and after MIST and DNA methylation. Emotional ratings are based on self-assessment mannikin (SAM) which is a non-verbal pictorial tool. Stress levels evaluated with a stress thermometer using a scale of 1-10; 1 indicating not at all, 10 very strong. Is there a mediating effect of DNA methylation on the correlation between subjective stress response and negative emotionality (e.g., internalizing symptoms and stress processing). Comparing pre-and post-pubertal girls
Correlation between DNA methylation and phsiological stress response | Measured once: 20 minutes for phsiological data during MRI measurement
  Correlation between HR, HRV and skin conductance changes during stress task (MIST) and DNA methylation. The interaction between physiological acute stress response and DNA methylation in relation to negative emotionality (e.g., internalizing symptoms and stress processing). Comparing pre-and post-pubertal girls
Correlation between DNA methylation and functional connectivity | Measured once with resting-state functional MRI, approximately 10 mintes
  The correlation between functional connectivity in brain networks (e.g., default mode network (DMN) and salience network (SN)) and DNA methlaytion. The correlation between regions of interest (i.e., amygdala, anterior cingulate cortex, and hippocampus) activity during rest condition and DNA methylation. Is there a mediating role of DNA methylation on the correlation between resting-state neuronal activity and negative emotionality (e.g., mood and anxiety symptoms)? Comparing pre- and post-pubertal girls.
Correlation between DNA methylation and brain gray matter structure | Measured once with MPRAGE MRI, approximately 10 minutes. Analyzed and reported over the course of the study, in average of 1 year
  The correlation between gray matter volumes obtained from anatomical T1-weighted images in regions of interest (i.e., amygdala, dorsolateral prefrontal cortex, putamen, anterior cingulate, hippocampus, ventral striatum) and DNA methylation. Is there a mediating role of DNA methylation on the correlation between region of interest gray matter volumes and negative emotionality (e.g., stress processing, mood and anxiety symptoms). Comparing pre- and post-pubescent girls.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Nieratschker, Prof., Principal Investigator — University Hospital Tuebingen; Mirac Nur Musaoglu, MD, Study Director — University Hospital Tuebingen
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy; Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study.
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.